CLINICAL TRIAL: NCT04696822
Title: Bioavailability Comparison of Epinephrine Following a Single Nasal Dose of Microspheres Powder With Epinephrine Intramuscular Injection in Adults With Seasonal Allergic Rhinitis With and Without Nasal Allergen Challenge
Brief Title: Bioavailability of Nasal Epinephrine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nasus Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NP-002
Record Dates: First submitted 2020-12-01; First posted 2021-01-06 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2021-10

CONDITIONS: Anaphylaxis
MeSH Terms: conditions — Anaphylaxis | interventions — Allergens; Epinephrine

STUDY DESIGN:
Intervention Model Description: Open-label, single-dose, two-period, three-treatment, fixed-sequence, comparative bioavailability study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adults with seasonal allergic rhinitis (Experimental): Single administration of 1.6mg or 3.2 mg Epinephrine powder nasal spray, with or without allergenic challenge, and single IM 0.3 mg Epinephrine without allergenic challenge.
  Interventions: Drug: Epinephrine Nasal Product, 1.6 mg; Drug: Epinephrine nasal product, 1.6 mg + allergen; Drug: Epinephrine Injection 0.3 mg; Drug: Epinephrine Nasal Product, 3.2 mg; Drug: Epinephrine Nasal Product, 3.2 mg + allergen

INTERVENTIONS:
Drug: Epinephrine Nasal Product, 1.6 mg — Single dose Nasal powder spray without allergen challenge
  Other Names: FMXIN002 Microspheres Powder
Drug: Epinephrine nasal product, 1.6 mg + allergen — Single dose Nasal powder spray with allergen challenge
  Other Names: FMXIN002 Microspheres Powder
Drug: Epinephrine Injection 0.3 mg — Intramuscular injection
  Other Names: EpiPen
Drug: Epinephrine Nasal Product, 3.2 mg — Twice dose Nasal powder spray without allergen challenge
  Other Names: FMXIN002 Microspheres Powder, double dose
Drug: Epinephrine Nasal Product, 3.2 mg + allergen — Twice dose Nasal powder spray with allergen challenge
  Other Names: FMXIN002 Microspheres Powder, double dose

SUMMARY:
A Study to Compare the Bioavailability of Epinephrine following a Single Nasal Dose of FMXIN002 Microspheres Powder with Epinephrine 0.3 mg Intramuscular Injection in Adult Subjects with Seasonal Allergic Rhinitis with and without Nasal Allergen Challenge

DETAILED DESCRIPTION:
Study Design: Open-label, single-dose, two-period, three-treatment, fixed-sequence, comparative bioavailability study Study Population: Non-smoking, male and female subjects, from 18 to 55 years of age with known history of hay fever, seasonal allergies, or rhinitis during the last year.

ELIGIBILITY:
Inclusion Criteria:

The following inclusion criteria will be assessed at screening (within 28 days prior to the first drug administration):

1. Non-smoking, male and female subjects from 18 to 55 years of age.
2. Documented Positive skin allergy test during the last year.
3. History of hay fever, seasonal allergies, or rhinitis.
4. BMI ≥18 and <=30 kg/m2.
5. Females may be of childbearing or non-childbearing potential:

   * Childbearing potential:

     o Physically capable of becoming pregnant
   * Non-childbearing potential:

     * Surgically sterile (i.e., both ovaries removed, uterus removed, or bilateral tubal ligation); and/or
     * Postmenopausal (no menstrual period for at least 12 consecutive months without any other medical cause.
6. Willing to use acceptable, effective methods of contraception.
7. Able to tolerate venipuncture.
8. Be informed of the nature of the study and give written consent prior to any study procedure.
9. Willing and being able to remain in the clinic for the entire duration of the confinement period.
10. Have good intravenous access on both arms and hands.

    -

    Exclusion Criteria:

    Known history or presence of clinically significant neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, genitourinary, psychiatric, or cardiovascular disease or any other condition which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.

    Known or suspected carcinoma. Known history or presence of hypersensitivity or idiosyncratic reaction to epinephrine, sulfite, other excipients of epinephrine auto-injector, or any other drug substances with similar activity.

    Known history or presence of clinically significant lactose, galactose, or fructose intolerance.

    Known history or presence of cardiac arrythmias, coronary artery disease or organic heart disease.

    Known history or presence of hyperthyroidism. Known history or presence of diabetes. Known history or presence of Parkinson's disease. Known history or presence of any food allergy. Presence of hepatic or renal dysfunction. Presence of nostril or septum piercing. Presence of abnormal nasal anatomy (e.g., polyps, unilateral or bilateral abnormalities of the nares, nasal turbinates, or septum including deviated septum).

    History of nasal surgery. Presence of a medical condition requiring regular medication (prescription and/or over-the-counter) with systemic absorption.

    History of drug or alcohol addiction requiring treatment or positive alcohol breath test at check-in.

    Any acute illness (e.g. cold, acute infection) which is considered significant by the Investigator and that has not resolved within 7 days before the first drug administration.

    Positive test result for HIV, Hepatitis B surface antigen, or Hepatitis C antibody.

    Positive test result for urine drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, opiates, phencyclidine, and tricyclic antidepressants) or urine cotinine.

    Difficulty fasting or consuming standard meals. Inability to communicate well with the Investigators and staff (e.g., language problem, poor mental development or impaired cerebral function).

    Non-cooperative or unwilling to sign consent form or unwilling to attend scheduled clinic visits and/or comply with the study protocol.

    Use of tobacco or nicotine-containing products within 6 months prior to drug administration.

    Females who:
    * Have discontinued or changed the use of implanted, intrauterine, intravaginal, or injected hormonal contraceptives within 6 months prior to drug administration;
    * Have discontinued or changed the use of oral or patch hormonal contraceptives within 1 month prior to drug administration;
    * Are pregnant (serum hCG consistent with pregnancy); or
    * Are lactating.

    Donation or loss of whole blood (including clinical trials):
    * ≥50 mL and <500 mL within 30 days prior to drug administration;
    * ≥500 mL within 56 days prior to drug administration. Participation in a clinical trial that involved administration of an investigational medicinal product within 30 days prior to drug administration, or recent participation in a clinical investigation that, in the opinion of the Investigator, would jeopardize subject safety or the integrity of the study results.

    On a special diet within 30 days prior to drug administration (e.g., liquid, protein, raw food diet).

    Have had a tattoo or body piercing within 30 days prior to drug administration. Have clinically significant findings in vital signs measurements at screening. Systolic blood pressure increase or decrease in value by more than 20 mmHg and/or diastolic blood pressure decrease in value by more than 10 mmHg, from supine or sitting to standing position during orthostatic blood pressure measurement taken at screening.

    Have clinically significant findings in a 12-lead ECG. Have clinically significant abnormal laboratory values and hemoglobin <135 g/L for males or <120 g/L for females at screening.

    Have significant diseases at the screening. Have clinically significant findings from a physical examination.

    Use of the following drugs within 14 days prior to drug administration:
    * Alpha-adrenergic blocking drugs (e.g., phentolamine);
    * Anti-arrhythmics;
    * Beta-adrenergic blocking drugs (e.g., propranolol);
    * Cardiac glycosides;
    * Diuretics;
    * Drugs having an effect on cytochrome P450 (CYP450);
    * Enzyme-altering drugs (e.g., barbiturates, phenothiazines, cimetidine, carbamazepine, etc.);
    * Enzyme-modifying drugs known to induce/inhibit hepatic drug metabolism;
    * Ergot alkaloids;
    * Levothyroxine sodium;
    * Monoamine oxidase inhibitors;
    * Oral or topical corticosteroids;
    * Phenylephrine;
    * Reserpine-type or clonidine-type antihypertensives;
    * Sodium cromoglycate; or
    * Tricyclic antidepressants.

    Use of the following drugs within 7 days prior to drug administration:
    * Nasal decongestants;
    * Nonsteroidal anti-inflammatory drugs (NSAIDs); or
    * Oral or topical antihistamines.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
Epinephrine in blood - Cmax | -1 hour to 8 hours post-dose
  pharmacokinetic analysis
Epinephrine in blood- Tmax | -1 hour to 8 hours post-dose
  pharmacokinetic analysis
Epinephrine in blood- AUC | -1 hour to 8 hours post-dose
  pharmacokinetic analysis
Epinephrine in blood- T half | -1 hour to 8 hours post-dose
  pharmacokinetic analysis

SECONDARY OUTCOMES:
body temperature | morning
  Safety Monitoring
Hemoglobin level in blood | at check-in morning
  Safety Monitoring, blood test
blood hematocrit | check-in morning
  Safety Monitoring: the ratio of the volume of red blood cells to the total volume of blood
Blood pressure | Prior to drug administration
  Vital signs
Pulse | Prior to drug administration
  Vital signs
Blood pressure | 15 minutes
  Vital signs
Pulse | 15 minutes
  Vital signs
Blood pressure | 30 minutes
  Vital signs
Pulse | 30 minutes
  Vital signs
Blood pressure | 45 minutes
  Vital signs
Pulse | 45 minutes
  Vital signs
Blood pressure | 1 hour
  Vital signs
Pulse | 1 hour
  Vital signs
Blood pressure | 2 hours
  Vital signs
Pulse | 2 hours
  Vital signs
Blood pressure | 4 hours post-dose
  Vital signs
Pulse | 4 hours post-dose
  Vital signs
electrocardiogram | 3 hours prior to drug administration
  Safety Monitoring
electrocardiogram | 45 minutes
  Safety Monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Yoseph Caraco, Prof., Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Ein Kerem, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tal Y, Ribak Y, Rubin L, Talmon A, Shamriz O, Hershko AY, Blotnick S, Bouhajib M, Krayz GT, Abrutzky C, Megiddo D, Lapidot T, Caraco Y. Fast Acting, Dry Powder, Needle-Free, Intranasal Epinephrine Spray: A Promising Future Treatment for Anaphylaxis. J Allergy Clin Immunol Pract. 2023 Oct;11(10):3047-3054. doi: 10.1016/j.jaip.2023.06.044. Epub 2023 Jun 30. PMID 37394178
- See also: full text open article — https://doi.org/10.1016/j.jaip.2023.06.044